CLINICAL TRIAL: NCT03683017
Title: OrthoPulse 2.0 and 2.1 Product Evaluation and Assessing Clinical Effectiveness: A Feasibility Study
Brief Title: OrthoPulse 2.0 and 2.1 Feasibility Evaluation
Acronym: BX13
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX13
Record Dates: First submitted 2018-02-27; First posted 2018-09-25 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Malocclusion
Keywords: Malocclusion; Photobiomodulation; Biolux; OrthoPulse; Low-level laser therapy; Orthodontics
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable; Orthodontic Appliances, Fixed; Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- I-OP2.0 (Experimental): Patients receive Invisalign orthodontic treatment, with 3.5 day Aligner changes, by the qualified Principal Investigator (PI). Patients receive OrthoPulse 2.0 device.
  Interventions: Device: OrthoPulse 2.0; Device: Invisalign 3.5 Day Wear
- I-OP2.1 (Experimental): Patients receive Invisalign orthodontic treatment, with 3.5 day Aligner changes, by the qualified Principal Investigator (PI). Patients receive OrthoPulse 2.1 device.
  Interventions: Device: OrthoPulse 2.1; Device: Invisalign 3.5 Day Wear
- F-OP2.0 (Experimental): Patients receive fixed appliance orthodontic treatment by the qualified Principal Investigator (PI). Patients receive OrthoPulse 2.0 device.
  Interventions: Device: OrthoPulse 2.0; Device: Fixed Orthodontic Appliances (Braces)

INTERVENTIONS:
Device: OrthoPulse 2.0 — Patients are given OrthoPulse 2.0, an extended OrthoPulse device with no zone control (ability for doctor to control treatment regions). Patients complete 10 minute treatments (5 minutes each arch) every day.
  Arms: F-OP2.0; I-OP2.0
Device: OrthoPulse 2.1 — Patients are given OrthoPulse 2.1, an extended OrthoPulse device with zone control (ability for doctor to control treatment regions). Patients complete 10 minute treatments (5 minutes each arch) every day.
  Arms: I-OP2.1
Device: Invisalign 3.5 Day Wear — Patients are are fitted with sets of clear orthodontic Aligners by a qualified Principal Investigator (PI) using a ClinCheck plan by Align Technology. Aligners are worn for approximately 22 hours a day, and switched every 3.5 days.
  Arms: I-OP2.0; I-OP2.1
Device: Fixed Orthodontic Appliances (Braces) — Patients are fitted with a set of brackets and wires, as per standard orthodontic treatment by a qualified Principal Investigator (PI).
  Arms: F-OP2.0

SUMMARY:
OrthoPulse is a device that uses near-infrared light therapy in order to decrease orthodontic treatment time. The aim of this study is to evaluate OrthoPulse products modified with extended arrays, OrthoPulse 2.0 and OrthoPulse 2.1, and to assess their clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent must be obtained before any assessment is performed
* Patient must be 11 years of age or older; minors will only be included in the study with the consent of the Parent/Legal Authorized Representative (LAR)
* Presence of permanent dentition
* Eligible and scheduled for full mouth fixed orthodontic treatment or Invisalign
* Good oral hygiene
* Likely to be compliant to OrthoPulse 2.0 and 2.1 use, aligner wear and elastic wear
* Have a compatible iOS or Android device and are willing to download the OrthoPulse app for frequent automatic syncing of use data

Exclusion Criteria:

* Patient is currently enrolled in another clinical study
* Periodontally involved teeth, acute oral infection or periodontal disease
* Use of bisphosphonates (osteoporosis drugs) during the study
* Use of drugs that may cause photosensitivity
* History of photosensitivity
* History of poor oral hygiene, per the discretion of the Principal Investigator (PI)
* Epilepsy
* Patient plans to relocate over the treatment period
* Smoker or use of any tobacco containing products per the discretion of the PI

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Feedback on general experience | Through Study Completion, approx. 2 years
  Assess doctor and patient feedback on the general experience with OrthoPulse 2.0 and OrthoPulse 2.1 as measured in the electronic data capture system.
Feedback on clinical performance | Through Study Completion, approx. 2 years
  Assess doctor subjective and objective feedback on the clinical performance of OrthoPulse 2.0 and OrthoPulse 2.1 as measured in the electronic data capture system.
Adverse events | Through Study Completion, approx. 2 years
  Confirm initial safety of OrthoPulse 2.0 and OrthoPulse 2.1

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brawn, DDS, Study Director — Biolux Research Holdings, Inc.
Locations (7):
- United States (6):
  - Dickerson Orthodontics, Chandler, Arizona
  - Dickerson Orthodontics, Peoria, Arizona
  - Dickerson Orthodontics, Phoenix, Arizona
  - Dickerson Orthodontics, Scottsdale, Arizona
  - Bella Smile, San Francisco, California
  - Chenin Orthodontics, Henderson, Nevada
- Sphinx Orthodontics, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482
- [Background] Yamaguchi M, Hayashi M, Fujita S, Yoshida T, Utsunomiya T, Yamamoto H, Kasai K. Low-energy laser irradiation facilitates the velocity of tooth movement and the expressions of matrix metalloproteinase-9, cathepsin K, and alpha(v) beta(3) integrin in rats. Eur J Orthod. 2010 Apr;32(2):131-9. doi: 10.1093/ejo/cjp078. Epub 2010 Feb 16. PMID 20159792
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Shaughnessy T, Kantarci A, Kau CH, Skrenes D, Skrenes S, Ma D. Intraoral photobiomodulation-induced orthodontic tooth alignment: a preliminary study. BMC Oral Health. 2016 Jan 13;16:3. doi: 10.1186/s12903-015-0159-7. PMID 26762247
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] Masha RT, Houreld NN, Abrahamse H. Low-intensity laser irradiation at 660 nm stimulates transcription of genes involved in the electron transport chain. Photomed Laser Surg. 2013 Feb;31(2):47-53. doi: 10.1089/pho.2012.3369. Epub 2012 Dec 16. PMID 23240874
- [Background] Dickerson TE. Invisalign with Photobiomodulation: Optimizing Tooth Movement and Treatment Efficacy with a Novel Self-Assessment Algorithm. J Clin Orthod. 2017 Mar;51(3):157-165. No abstract available. PMID 28646819
- [Background] Arany PR. Craniofacial Wound Healing with Photobiomodulation Therapy: New Insights and Current Challenges. J Dent Res. 2016 Aug;95(9):977-84. doi: 10.1177/0022034516648939. Epub 2016 May 9. PMID 27161014
- [Background] Ojima K, Dan C, Kumagai Y, Schupp W. Invisalign Treatment Accelerated by Photobiomodulation. J Clin Orthod. 2016 May;50(5):309-17; quiz 319-20. No abstract available. PMID 27323274
- [Background] Shaughnessy TG. Long-Distance Orthodontic Treatment with Adjunctive Light Therapy. J Clin Orthod. 2015 Dec;49(12):757-69. No abstract available. PMID 26799997
- [Background] Guo J, Wang Q, Wai D, Zhang QZ, Shi SH, Le AD, Shi ST, Yen SL. Visible red and infrared light alters gene expression in human marrow stromal fibroblast cells. Orthod Craniofac Res. 2015 Apr;18 Suppl 1(0 1):50-61. doi: 10.1111/ocr.12081. PMID 25865533